CLINICAL TRIAL: NCT02910258
Title: Etude de l'efficacité et de la tolérance de l'interféron-pégylé Dans Les myélofibroses
Brief Title: Interferon-pegyle α2a Efficiency and Tolerance in Myelofibrosis
Acronym: PEG-MF
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PEG-MF
Record Dates: First submitted 2016-08-26; First posted 2016-09-22 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Myelofibrosis
Keywords: myelofibrosis; pegylated interferon
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients who carried primary or secondary myelofibrosis from Philadelphia negative MPNs (PMF/SMF) and who are treated or are about to be treated with pegylated-interferon (mostly α2a) are eligible to this prospective study. Biological and clinical parameters will be collected from the beginning of the drug use until last news.

A non-opposition consent form need to be signed before entering this study.

DETAILED DESCRIPTION:
In all centres interested, patients who were diagnosed for PMF/SMF can be treated with oral or sub-cutaneous drugs in order to reduce clinical symptoms and biological abnormalities belonging to these diseases.

Pegylated-interferon is one of the better weapons that can be used in these cases. These treatments are well known and used from many years in french hematological centres.

The investigators to collect clinical and biological data from patients treated with pegylated-interferon α2a (the most use) in case of PMF/SMF in order to assess efficacity and tolerance to this drug. The prescription of the product and the dose are under the responsibility of each practician.

Clinical data collected: disease and patients characteristics at the time of diagnosis and at the beginning of the drug use, spleen and liver size, presence of constitutive symptoms, transfusion needs.

Biological data collected: complete hemogram, CD34+ cells count, allele burden of JAK2V617F and calreticulin clones if DNA samples are collected.

These data will be collected avery 3 months during the two first years and every 6 months after.

The investigators also recorded adverse side effects if significative, the concomitant use of hematological drugs (cytoreductive treatments, ASE...), modalities of prescription of the drugs and the reason for stopping the drug and etiology of death if happened.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary Myelofibrosis
* Prescription of pegylated interferon α2a
* Age > 18 years-old

Exclusion Criteria:

* Other MPNs treated with pegylated interferon α2a
* Patients treated for PMF or SMF but without pegylated interferon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed for PMF or SMF and treated with pegykated interferon α2a
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2012-09; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Efficiency of the interferon in Myelofibrosis | Evaluation at 1 year
  Evaluation on the presence or not of splenomegaly and physical signs or the normalization of blood counts.

SECONDARY OUTCOMES:
Rate of survival of patients with Myelofibrosis under interferon | Evaluation at 5 years
  Patients dead or alive at this time
Tolerance of Interferon | Evaluation at 1 year
  Presence or not of psychiatric symptoms, cramps, hepatitic abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Ianotto, MD, Study Director — CHRU de Brest
Locations (12):
- France (12):
  - CHU d'Angers, Angers
  - Hopital du genevois, Annecy
  - CHRU de Brest, Brest
  - Centre Hospitalier du Mans, Le Mans
  - Centre Hospitalier de Lens, Lens
  - Institut Paoli Calmette, Marseille
  - CH des pays de Morlaix, Morlaix
  - Centre Hospitalier de Nice, Nice
  - AP-HP Hôpital Saint Louis, Paris
  - CHIC de Cornouaille, Quimper
  - Centre Hospitalier de Tours, Tours
  - CHU de Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ianotto JC, Chauveau A, Boyer-Perrard F, Gyan E, Laribi K, Cony-Makhoul P, Demory JL, de Renzis B, Dosquet C, Rey J, Roy L, Dupriez B, Knoops L, Legros L, Malou M, Hutin P, Ranta D, Benbrahim O, Ugo V, Lippert E, Kiladjian JJ. Benefits and pitfalls of pegylated interferon-alpha2a therapy in patients with myeloproliferative neoplasm-associated myelofibrosis: a French Intergroup of Myeloproliferative neoplasms (FIM) study. Haematologica. 2018 Mar;103(3):438-446. doi: 10.3324/haematol.2017.181297. Epub 2017 Dec 7. PMID 29217781